CLINICAL TRIAL: NCT04523480
Title: Randomized Control Trial of Long Acting Subcutaneous Testosterone Pellets for Hypogonadism: Testopel ® vs. Generic Testosterone Pellets.
Brief Title: Testopel ® vs. Generic Testosterone Pellets.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Empower Research Inc (Industry)
Responsible Party: Principal Investigator, Ranjith Ramasamy, MD, Director of Male Fertility and Andrology, University of Miami, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRBSITE00000555; 20192539 (Other: Western Institutional Review Board® (WIRB®))
Record Dates: First submitted 2020-08-11; First posted 2020-08-21 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Hypogonadism
Keywords: Low T; Low Testosterone
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Testopel 75mg Group (Experimental): Participants in this group will receive a one-time subcutaneous testosterone insertion of 10 x 75 mg pellets of Testopel for a total of 750 mg Testopel.
  Interventions: Drug: Testopel 75mg Drug Implant
- Compounded testosterone pellets 100mg Group (Active Comparator): Participants in this group will receive a one-time subcutaneous testosterone insertion of 8 x 100 mg compounded testosterone for a total of 800 mg compounded testosterone.
  Interventions: Drug: Testopel 100mg Drug Implant
- Compounded Testosterone pellets 200mg Group (Active Comparator): Participants in this group will receive a one-time subcutaneous testosterone insertion of 4 x 200 mg compounded testosterone for a total of 800 mg compounded testosterone.
  Interventions: Drug: Testopel 200mg Drug Implant

INTERVENTIONS:
Drug: Testopel 75mg Drug Implant — 75 mg Testosterone pellets administered subcutaneously.
  Arms: Testopel 75mg Group
Drug: Testopel 100mg Drug Implant — 100 mg Testosterone pellets administered subcutaneously.
  Arms: Compounded testosterone pellets 100mg Group
Drug: Testopel 200mg Drug Implant — 200 mg Testosterone pellets administered subcutaneously.
  Arms: Compounded Testosterone pellets 200mg Group

SUMMARY:
The purpose of this study is to evaluate changes in vascular parameters in subjects receiving Testopel 75mg (one time) versus subjects receiving Compounded Testosterone pellets 100mg (one time) versus subjects receiving Compounded Testosterone pellets 200mg (one time) to participant with clinical hypogonadism.

DETAILED DESCRIPTION:
Hypogonadism, or low testosterone (Low T), is the deficiency in producing testosterone by the testes. Testosterone pellets is a long-acting formulation of Testosterone Replacement Therapy (TRT) that is delivered subcutaneously to men diagnosed with low T. Advantages to subcutaneous testosterone pellets include ease of delivery and decreased risk of the medication being transfer upon skin contact to woman or children. Long acting testosterone replacement Implantation of six to ≥10 testosterone pellets (450 to ≥750 mg) increased total testosterone into the therapeutic range at 1 month post-implantation and sustained therapeutic levels (>300) for 4-6 months.

Participants will be randomly assigned to 1 of 3 study groups. In one of the groups the treatment will include implantation of Testopel ® 750mg (10 pellets with 75mg pellet) one time, in the second group, treatment will include compounded subcutaneous testosterone 800mg (8 pellets with 100mg pellet) one time and in the third group, treatment will include compounded subcutaneous testosterone 800mg (4 pellets with 200mg pellet) one time.

The treatment takes approximately 30 minutes and will include: Clean and numb the insertion site with lidocaine at 1%, followed by small incision in the skin, implantation of pellets into subdermal fat layer and sealing the incision with Steri-strip. This is the current standard of care of Testopel insertion and same procedure will be followed with both compounded and commercial pellets.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign and date the study consent form(s), which have been approved by an Institutional Review Board (IRB). Written consent must be obtained prior to the initiation of any study procedures.
* Male between 18 and 75 years of age.
* Documented diagnosis of primary hypogonadism (congenital or acquired) or hypogonadotropic hypogonadism (congenital or acquired).
* Serum total testosterone < 300 ng/dL on 2 measurements
* Naïve to androgen replacement or has discontinued current treatment and completed a washout of 4 weeks following androgen treatment.
* Judged to be in good general health as determined by the principal investigator based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* History of significant sensitivity or allergy to androgens, or product excipients.
* Clinically significant findings in the pre-study examinations including abnormal breast examination requiring follow-up, abnormal ECG.
* Abnormal prostate digital rectal examination (DRE) with palpable nodule(s) or International Prostate Symptom Score (I-PSS) score > 19 points.
* Body mass index (BMI) ≥ 40 kg/m2.
* Clinically significant abnormal laboratory value, in the opinion of the investigator, in serum chemistry, hematology, or urinalysis including but not limited to:

  1. Baseline hemoglobin > 16 g/dL
  2. Hematocrit < 35% or > 50%
  3. prostate-specific antigen (PSA) > 4 ng/mL
* History of seizures or convulsions, including febrile, alcohol or drug withdrawal seizures.
* History of any clinically significant illness, infection, or surgical procedure within 4 weeks prior to study drug administration.
* History of stroke or myocardial infarction within the past 5 years.
* History of, or current or suspected, prostate or breast cancer.
* History of diagnosed, severe, untreated, obstructive sleep apnea.
* History of abuse of alcohol or any drug substance in the opinion of the investigator within the previous 2 years.
* Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 12 weeks prior to the start of treatment.
* Inadequate venous access for collection of serial blood samples required for pharmacokinetic profiles.
* Receipt of any investigational product within 4 weeks or within 5 half-lives prior to the start of treatment.
* Inability to understand and provide written informed consent for the study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjith Ramasamy, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Department of Urology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corona G, Rastrelli G, Maggi M. Diagnosis and treatment of late-onset hypogonadism: systematic review and meta-analysis of TRT outcomes. Best Pract Res Clin Endocrinol Metab. 2013 Aug;27(4):557-79. doi: 10.1016/j.beem.2013.05.002. Epub 2013 Jul 5. PMID 24054931
- [Background] Walker WH. Testosterone signaling and the regulation of spermatogenesis. Spermatogenesis. 2011 Apr;1(2):116-120. doi: 10.4161/spmg.1.2.16956. PMID 22319659
- [Background] Katznelson L, Finkelstein JS, Schoenfeld DA, Rosenthal DI, Anderson EJ, Klibanski A. Increase in bone density and lean body mass during testosterone administration in men with acquired hypogonadism. J Clin Endocrinol Metab. 1996 Dec;81(12):4358-65. doi: 10.1210/jcem.81.12.8954042.
- [Background] Finkelstein JS, Klibanski A, Neer RM, Greenspan SL, Rosenthal DI, Crowley WF Jr. Osteoporosis in men with idiopathic hypogonadotropic hypogonadism. Ann Intern Med. 1987 Mar;106(3):354-61. doi: 10.7326/0003-4819-106-3-. PMID 3544993
- [Background] Jockenhovel F, Vogel E, Reinhardt W, Reinwein D. Effects of various modes of androgen substitution therapy on erythropoiesis. Eur J Med Res. 1997 Jul 28;2(7):293-8. PMID 9233903
- [Background] Behre HM, Bohmeyer J, Nieschlag E. Prostate volume in testosterone-treated and untreated hypogonadal men in comparison to age-matched normal controls. Clin Endocrinol (Oxf). 1994 Mar;40(3):341-9. doi: 10.1111/j.1365-2265.1994.tb03929.x. PMID 7514512
- [Background] Davidson JM, Camargo CA, Smith ER. Effects of androgen on sexual behavior in hypogonadal men. J Clin Endocrinol Metab. 1979 Jun;48(6):955-8. doi: 10.1210/jcem-48-6-955. PMID 447801
- [Background] Snyder PJ, Peachey H, Berlin JA, Hannoush P, Haddad G, Dlewati A, Santanna J, Loh L, Lenrow DA, Holmes JH, Kapoor SC, Atkinson LE, Strom BL. Effects of testosterone replacement in hypogonadal men. J Clin Endocrinol Metab. 2000 Aug;85(8):2670-7. doi: 10.1210/jcem.85.8.6731. PMID 10946864
- [Background] Baillargeon J, Urban RJ, Ottenbacher KJ, Pierson KS, Goodwin JS. Trends in androgen prescribing in the United States, 2001 to 2011. JAMA Intern Med. 2013 Aug 12;173(15):1465-6. doi: 10.1001/jamainternmed.2013.6895. No abstract available. PMID 23939517
- [Background] Ullah MI, Riche DM, Koch CA. Transdermal testosterone replacement therapy in men. Drug Des Devel Ther. 2014 Jan 9;8:101-12. doi: 10.2147/DDDT.S43475. eCollection 2014. PMID 24470750

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Testopel 75mg Group | Compounded Testosterone Pellets 100mg Group | Compounded Testosterone Pellets 200mg Group
Started | 33 | 42 | 0
Completed | 3 | 7 | 0
Not Completed | 30 | 35 | 0
Not completed — Lost to Follow-up | 30 | 35 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled to the 200mg group due to complications with the compounding pharmacies ability to produce the medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Testopel 75mg Group | Compounded Testosterone Pellets 100mg Group | Compounded Testosterone Pellets 200mg Group | Total
Number analyzed (Participants) | 33 | 42 | 0 | 75
Age, Continuous [Median (Full Range); unit: years] | 54.5 [35 to 74] | 52.5 [22 to 69] |  | 53.5 [22 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 33 | 42 | 0 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 29 | 0 | 53
  Not Hispanic or Latino | 9 | 13 | 0 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 6 | 0 | 9
  White | 6 | 7 | 0 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 24 | 29 | 0 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change in Testosterone (T) Levels
Description: Changes in serum Testosterone levels are assessed in ng/dL
Time Frame: Baseline, 2 months, 4 months, and 6 months
Population: Zero participants were enrolled into the "Compounded Testosterone pellets 200mg Group" due to the pharmacy being unable to produce the investigational product at that dosage amount.
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | Testopel 75mg Group | Compounded Testosterone Pellets 100mg Group | Compounded Testosterone Pellets 200mg Group
Number analyzed (Participants) | 33 | 42 | 0
ng/dL
  Baseline | 219.5 [194 to 252] | 202.3 [143.5 to 256] |
  Month 2 | 543 [460 to 716.5] | 696.5 [591 to 822] |
  Month 4 | 290 [209 to 439] | 277 [228 to 378] |
  Month 6 | 209 [155 to 267] | 241 [158 to 287] |

2. Secondary Outcome: Change in Hematocrit (Hct) Levels.
Description: Changes in serum Hct levels are assessed in %.
Time Frame: Baseline, 2 months, 4 months, and 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hematocrit percentage
Arm/Group | Testopel 75mg Group | Compounded Testosterone Pellets 100mg Group | Compounded Testosterone Pellets 200mg Group
Number analyzed (Participants) | 33 | 42 | 0
hematocrit percentage
  Baseline | 43.7 [42.3 to 46.7] | 42.8 [39.3 to 45.6] |
  Month 2 | 46.1 [42.4 to 49.4] | 46.7 [42.1 to 48.4] |
  Month 4 | 45.9 [42.8 to 48.7] | 45.8 [44.4 to 46.8] |
  Month 6 | 46 [43.1 to 47.3] | 43 [40.8 to 46.7] |

3. Secondary Outcome: Change in PSA Levels
Description: Change in serum Prostate Specific Antigen (PSA) levels are assessed in ng/mL.
Time Frame: Baseline, 2 months, 4 months, and 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Testopel 75mg Group | Compounded Testosterone Pellets 100mg Group | Compounded Testosterone Pellets 200mg Group
Number analyzed (Participants) | 33 | 42 | 0
ng/mL
  Baseline | 0.9 [0.5 to 1.6] | 0.4 [0.3 to 0.8] |
  Month 2 | 1.1 [0.6 to 1.85] | 0.75 [0.5 to 1.2] |
  Month 4 | 1 [0.5 to 1.6] | 0.65 [0.5 to 1.2] |
  Month 6 | 0.8 [0.6 to 1.7] | 0.5 [0.3 to 0.6] |

4. Secondary Outcome: Change in Estradiol Levels
Description: Change in serum estradiol levels are assessed in pg/mL.
Time Frame: Baseline, 2 months, 4 months, and 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Testopel 75mg Group | Compounded Testosterone Pellets 100mg Group | Compounded Testosterone Pellets 200mg Group
Number analyzed (Participants) | 33 | 42 | 0
pg/mL
  Baseline | 18.2 [8.5 to 25] | 20.6 [8.5 to 24.3] |
  Month 2 | 29.1 [21.3 to 35.4] | 42.7 [42.1 to 48.4] |
  Month 4 | 13.7 [8.1 to 24.6] | 18.4 [6.9 to 29.6] |
  Month 6 | 14.3 [0.1 to 17.6] | 18.8 [7 to 22.7] |

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated after implantation, and at each follow up visit (months 2, 4, and 6).
Description: zero subjects were enrolled to the 200mg treatment arm.
Arm/Group | Testopel 75mg Group | Compounded Testosterone Pellets 100mg Group | Compounded Testosterone Pellets 200mg Group
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/42 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/42 | 0/0
Other Adverse Events (participants affected / at risk) | 1/33 | 0/42 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testopel 75mg Group (N=33) | Compounded Testosterone Pellets 100mg Group (N=42) | Compounded Testosterone Pellets 200mg Group (N=0)
Pellet Extrusion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT04523480/Prot_SAP_000.pdf